CLINICAL TRIAL: NCT00514098
Title: An Observational Cohort Study of Women Following HIV-1 Seroconversion in Microbicide Trials
Brief Title: Observational Study of HIV Infected Women Previously Enrolled in Other Microbicide Trials
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-015; 5UM1AI068633 (NIH); 10529 (Other Grant/Funding Number: DAIDS Protocol ID)
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: HIV Infections
Keywords: Microbicide; Seroconversion; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine collection, pelvic, vaginal, and cervicovaginal sampling
Oversight: Data Monitoring Committee: No

SUMMARY:
A new approach to HIV prevention currently being studied includes the use of topical microbicides and orally administered anti-HIV drugs. The purpose of this study is to better understand the impact of microbicides in women who are diagnosed with HIV-1 during participation in previous microbicide trials.

DETAILED DESCRIPTION:
It is necessary to monitor HIV over long periods of time in order to better understand the impact of microbicides and anti-HIV drugs on the progression of HIV infection in those who become infected or are unknowingly already infected while receiving these drugs. The purpose of this study is to determine the effects of microbicides or oral anti-HIV drugs over time in HIV infected women who were previously enrolled in other microbicide trials.

The study will remain open to accrual for the duration of MTN funding, and will use two follow-up visit schedules, one based on the date of diagnosis in the parent study, and one based on the initiation of antiretroviral treatment (ART). Participants who have not initiated ART at the time of enrollment in this study will follow the schedule based on the date of diagnosis. Participants who have already begun ART at the time of enrollment will follow the schedule based on the date of ART initiation. Individuals enrolled with a starting date based on the date of ART initiation will have their first follow-up visit at Week 2 before resuming the rest of the schedule. On both schedules, follow-up visits occur at Months 1, 3, and 6 and every 6 months thereafter. Interim visits may be performed at any time during follow-up, and participants will be asked to attend a final study visit prior to their termination from the study. Participants may enroll any time after their HIV diagnosis and can leave the study at any time.

A physical exam; medical and medication history assessment; blood and urine collection; and pelvic, cervicovaginal lavage, and vaginal swab sampling will occur at all visits. A behavioral assessment will occur at select visits, and adherence and social harms assessments will occur at most visits. Sexually transmitted infection risk reduction/contraception and HIV-1 secondary counseling will occur at most visits. In addition, condoms will be provided at all visits to reduce further HIV transmission. ART will not be provided by this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV-1 infection during participation in any Microbicide Trials Network (MTN) clinical trial (including HPTN 035 and HPTN 059), according to the HIV testing algorithm of the parent MTN trial
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, makes participation in the study unsafe or interferes with the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who are diagnosed with HIV-1 during participation in previous microbicide trials
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2008-08-25 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HIV disease progression comparison | 12 months
  To compare HIV disease progression 12 months post seroconversion among participants assigned to an active agent compared to placebo/control participants.

SECONDARY OUTCOMES:
HIV disease progression comparison | Total duration of follow up
  To compare virologic and immunologic responses following initiation of antiretroviral therapy among participants assigned to an active agent versus placebo/control participants.
Virologic and immunologic response comparison | Total duration of follow up
  To compare virologic and immunologic responses following initiation of antiretroviral therapy among participants assigned to an active agent versus placebo/control participants.
HIV-1 drug resistance profile comparison | Total duration of follow up
  To compare the HIV-1 drug resistance profile, among antiretroviral therapy recipients at the time of virologic failure in participants assigned to an active agent versus placebo/control participants.
Sexual behavior and partnership status changes | Total duration of follow up
  To describe post seroconversion changes in sexual behaviors and partnership status of participants.

OTHER OUTCOMES:
HIV-1 drug resistance mutation evaluation | Total duration of follow up
  To evaluate the prevalence and persistence of HIV-1 drug resistance mutations in plasma and/or genital tract specimens after HIV-1 seroconversion using both standard and sensitive methods in specific subgroups of seroconverters.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Riddler, MD, Study Chair — University of Pittsburgh
Locations (18):
- Malawi (2):
  - College of Med. JHU CRS, Blantyre
  - University of North Carolina Lilongwe, Lilongwe
- South Africa (11):
  - Wits Reproductive Health Institute (WRHI), Johannesburg, Gauteng
  - CAPRISA- The Aurum Institute, Johannesburg, Guateng
  - Botha's Hill CRS, Durban, KwaZulu-Natal
  - CAPRISA eThewkini, Durban, KwaZulu-Natal
  - Overport CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Durban, KwaZulu-Natal
  - Verulam CRS, Durban, KwaZulu-Natal
  - South African Medical Research Council, Tongaat, Durban, KwaZulu-Natal
  - Umkomaas CRS, Durban, KwaZulu-Natal
  - Perinatal HIV Research Unit (HPRU), Johannesburg, Soweto
  - R. K. Khan CRS, Durban
- Makerere University- JHU Research Collaboration {MUJHU CARE LTD} CRS, Kampala, Uganda
- Kamwala Clinic CRS, Kamwala, Zambia
- Zimbabwe (3):
  - UZ-UCSF HIV Prevention Trials Unit, Harare, Chitungwiza
  - Seke South CRS, Chitungwiza
  - Spilhaus CRS, Harare

REFERENCES:
- [Result] Riddler SA, Balkus JE, Parikh UM, Mellors JW, Akello C, Dadabhai S, Mhlanga F, Ramjee G, Mayo AJ, Livant E, Heaps AL, O'Rourke C, Baeten JM; MTN-015 and MTN-020/ASPIRE Study Teams. Clinical and Virologic Outcomes Following Initiation of Antiretroviral Therapy Among Seroconverters in the Microbicide Trials Network-020 Phase III Trial of the Dapivirine Vaginal Ring. Clin Infect Dis. 2019 Jul 18;69(3):523-529. doi: 10.1093/cid/ciy909. PMID 30346511
- [Result] Riddler SA, Husnik M, Ramjee G, Premrajh A, Tutshana BO, Pather A, Siva S, Jeenarain N, Nair G, Selepe P, Kabwigu S, Palanee-Phillips T, Panchia R, Mhlanga F, Levy L, Livant E, Patterson K, Elharrar V, Balkus J. HIV disease progression among women following seroconversion during a tenofovir-based HIV prevention trial. PLoS One. 2017 Jun 28;12(6):e0178594. doi: 10.1371/journal.pone.0178594. eCollection 2017. PMID 28658251
- [Result] Riddler SA, Husnik M, Gorbach PM, Levy L, Parikh U, Livant E, Pather A, Makanani B, Muhlanga F, Kasaro M, Martinson F, Elharrar V, Balkus JE; MTN-015 Protocol Team for the Microbicide Trials Network. Long-term follow-up of HIV seroconverters in microbicide trials - rationale, study design, and challenges in MTN-015. HIV Clin Trials. 2016 Sep;17(5):204-11. doi: 10.1080/15284336.2016.1212561. Epub 2016 Jul 28. PMID 27465646